CLINICAL TRIAL: NCT07353775
Title: Intracardiac Echocardiography-Guided Cavotricuspid Isthmus Ablation With a Circular-Shaped Pulsed Field Ablation Catheter: A Prospective Study on Effectiveness and Safety
Brief Title: Intracardiac Echocardiography-Guided Cavotricuspid Isthmus Ablation With a Circular-Shaped Pulsed Field Ablation Catheter
Status: Recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PFA-CTI ablation
Record Dates: First submitted 2025-08-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF); Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Desmoglein 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: ICE-guided CTI ablation with PFA — Cavotricuspid isthmus ablation with a circular-shaped pulsed field ablation catheter guided by intracardiac echocardiography

SUMMARY:
This observational study aims to evaluate the effectiveness and safety of a circular-shaped pulsed field ablation (PFA) catheter for CTI ablation under the guidance of intracardiac echocardiography (ICE). The main question it aims to answer is:

Is the circular-shaped PFA catheter an effective and safe tool for achieving acute success for CTI ablation? Patients undergoing CTI ablation with a circular-shaped PFA catheter will be prospectively enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or persistent atrial fibrillation
* Aged 18 years or older
* Scheduled for CTI ablation
* Able and willing to provide written informed consent

Exclusion Criteria:

* Previous CTI ablation
* Significant congenital heart disease or structural anomaly affecting the CTI
* Active intracardiac thrombus
* Pregnancy or lactation
* Severe renal/hepatic insufficiency
* Active systemic infection or sepsis
* Life expectancy of less than 12 months
* Unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients scheduled for CTI ablation at Beijing Anzhen Hospital will be asked to participate in this study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Acute Success of CTI Block | Within the ablation procedure
  Bidirectional block was assessed immediately after the last ablation application and re-confirmed at the end of the 20-minute observation period.

SECONDARY OUTCOMES:
CTI Procedural Time | Within the ablation procedure
Total PF Application Time | Within the ablation procedure
Number of PFA Applications | Within the ablation procedure
Procedure-related Complications | Within 30 days after the ablation procedure
  Including vascular complications, cardiac tamponade, thromboembolic events, conduction system injury, or other adverse events judged procedure-related.
Freedom from Any Atrial Arrhythmia | 12 months
  Arrhythmia recurrence is defined as any documented atrial tachyarrhythmia (atrial flutter, atrial fibrillation, or atrial tachycardia) lasting ≥30 seconds, confirmed by ECG or ambulatory monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, China